CLINICAL TRIAL: NCT02892071
Title: Tri-split Face Study of Skin Resurfacing Modalities for the Treatment of Melasma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Our fellow completed the program before we were able to start the study
Sponsor: SUZAN OBAGI (Other)
Responsible Party: Sponsor-Investigator, SUZAN OBAGI, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO15090113
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- 22% TCA peel (Active Comparator): 22% trichloroacetic acid medium depth chemical peel applied to one of the three facial areas (based on random assignment- forehead, left cheek, right cheek)
  Interventions: Drug: 22% TCA peel
- CO2 laser (Active Comparator): CO2 ablative fractional laser resurfacing applied to one of the three facial areas (based on random assignment- forehead, left cheek, right cheek)
  Interventions: Device: CO2 laser
- Qs-NdYAG laser (Active Comparator): Long pulsed Q-switched Nd:Yag laser will be applied to one of the three facial areas (based on random assignment- forehead, left cheek, right cheek), performed at 2-week intervals for six sessions.
  Interventions: Device: Qs-NdYag laser

INTERVENTIONS:
Drug: 22% TCA peel — One of the three facial areas (based on random assignment- forehead, left cheek, right cheek) will be treated with one treatment with a 22% TCA Blue Peel, to achieve a level 2 frost (medium depth peel). Each treatment will take about 20 minutes. A 22% TCA concentration will be created by combining 5.5 mL of 30% TCA (from a purchased commercial bottle) with 2mL of blue dye (commercial), immediately before application.
  Other Names: medium depth chemical peel; TCA peel
  Arms: 22% TCA peel
Device: CO2 laser — One of the three facial areas (based on random assignment- forehead, left cheek, right cheek) will receive one treatment with one pass of the fractionated ablative 10,600 nm CO2 (CO2RE Laser, Syneron) at Core 70 mJ, Ring 50mJ, 40% coverage, 1 pass, 8 mm square pattern. Each treatment will take about 20 minutes.
  Other Names: CO2RE laser, ablative fractional laser
  Arms: CO2 laser
Device: Qs-NdYag laser — Long pulsed Q-switched Nd:Yag laser. One of the three facial areas (based on random assignment- forehead, left cheek, right cheek) will be treated with Q-switched (Qs) 1064 Nd:YAG (Medlite C3; 6 mm spot size, collimated homogenous flat- top beam profile, energy fluence 2.0 J/cm2, 5Hz), with 5% coverage and 2 passes (or until mild erythema detected). Treatments will be performed at 2-week intervals for six sessions. Each treatment will take about 20 minutes.
  Arms: Qs-NdYAG laser

SUMMARY:
Tri-split face study of skin resurfacing modalities for the treatment of melasma, comparing the medium depth trichloroacetic acid peel, CO2 laser and Qs-NdYag laser.

DETAILED DESCRIPTION:
Melasma is an acquired chronic and relapsing hyperpigmentation disorder, with a significant negative impact on the quality of life of patients. Melasma is more common in patients with skin of color and has also been linked to chronic ultraviolet (UV) and heat exposure, family history and hormonal factors. There are several studies in the literature using various therapies for melasma, including sun protection, topical therapies, lasers and chemical peels. However, many of these studies vary greatly in their efficacies and side effect profiles, due to varying and undelineated pre and post-op procedure regimens. Side effects of post-inflammatory hyper and hypopigmentation and rebound are reported in these studies. The investigators would like to conduct a tri-split face study that compares a 22% trichloroacetic acid (TCA) deep medium peel with an ablative fractionated CO2 laser and more pigment selective Q-switched (Qs) Nd:YAG laser. To minimize possible post-procedure side effects and melasma rebound, the investigators will perform above treatments in conjunction with an optimal skincare regimen, starting 6 weeks before and continuing after the treatments. The investigators will perform the 22% TCA chemical peel, CO2 laser and Qs-Nd:YAG at 6 weeks after the start of the skincare regimen, and repeat treatments with Qs-Nd:YAG at weeks 8, 10, and 12. The investigators will assess participants using standardized photos in conjunction with UV imaging (Visia CR) at weeks 0, 6, 16, 20 and 24 (6 months), by measuring the modified melasma area and severity index (mMASI) scores and visual analog scale (VAS) scores as graded by participants as well as by blinded physicians based on photos and UV imaging.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants
* 20 to 60 years old
* participants with melasma on forehead and both cheeks
* participants who failed topical therapy for melasma
* participants who have never tried other therapies for melasma

Exclusion Criteria:

* pregnancy
* lactation
* use of oral contraceptive (OCP) within 3 months of starting the study
* hormonal therapy within 3 months of starting the study
* hormonal intrauterine device (IUD) within 3 months of starting the study
* history of poor wound healing or abnormal scarring
* history of lip or face herpes simplex virus infections
* active facial skin infection
* history of connective tissue disorders (such as lupus or scleroderma)
* history of isotretinoin therapy within 6 months of starting the study
* history of chemical peels, dermabrasion, laser therapy or intense pulse light (IPL) within 6 months before enrollment into the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
modified melasma area and severity index (mMASI) score | 6 months
  score calculated by measuring darkness of pigment of melasma patch area

SECONDARY OUTCOMES:
visual analog scale (VAS) assessment by physicians | 6 months
  CR

OTHER OUTCOMES:
participant satisfaction assessment | 6 months
  Participants will score their satisfaction with improvement for each modality

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Obagi, MD, Principal Investigator — University of Pittsburgh Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moubasher AE, Youssef EM, Abou-Taleb DA. Q-switched Nd: YAG laser versus trichloroacetic acid peeling in the treatment of melasma among Egyptian patients. Dermatol Surg. 2014 Aug;40(8):874-82. doi: 10.1097/DSS.0000000000000065. PMID 25068546
- [Result] Trelles MA, Velez M, Gold MH. The treatment of melasma with topical creams alone, CO2 fractional ablative resurfacing alone, or a combination of the two: a comparative study. J Drugs Dermatol. 2010 Apr;9(4):315-22. PMID 20514787
- [Result] Jalaly NY, Valizadeh N, Barikbin B, Yousefi M. Low-power fractional CO(2) laser versus low-fluence Q-switch 1,064 nm Nd:YAG laser for treatment of melasma: a randomized, controlled, split-face study. Am J Clin Dermatol. 2014 Aug;15(4):357-63. doi: 10.1007/s40257-014-0080-x. PMID 24858737